CLINICAL TRIAL: NCT05465629
Title: Testing the Efficacy of Viome-designed Condition-based Supplements and Viome Precision Supplements to Improve Clinical Outcomes for Gastrointestinal Conditions
Brief Title: Viome Nutritional Programs to Improve Clinical Outcomes for Gastrointestinal Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V211.1
Record Dates: First submitted 2022-07-08; First posted 2022-07-20 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Health
Keywords: Nausea; Vomiting; Diarrhea; Constipation; Bloating; Gastroesophageal; Viome; Nutrition; Supplements; VPNP; Viome precision nutrition program; Reflux; Diet; Microbiome; Biome; Gastrointestinal
MeSH Terms: conditions — Nausea; Vomiting; Diarrhea; Constipation; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, cohort study divided into three arms: 1) control group (placebo), 2) condition-based supplement, 3) precision-supplement
Who Masked: Participant
Masking Description: Once enrolled, participants are randomized into one of the three arms. The coded supplements with blinded labels are shipped to the participants. The participants are not aware of which group they are randomized into.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (No Intervention): Participants who have gastrointestinal issues are randomized into this arm. They may be provided with any combination of nutritional recommendations and supplements. Placebo capsules will contain inert and inactive materials. Participants may need to use a mobile app in order to participate in the trial.
- Viome's Precision Nutrition Program (Active Comparator): Participants who have gastrointestinal issues are randomized into this arm. They may be provided with any combination of nutritional recommendations and supplements. Participants may need to use a mobile app in order to participate in the trial.
  Interventions: Combination Product: VIOME Precision Nutrition Program
- Viome's condition-based supplements (Active Comparator): Participants who have gastrointestinal issues are randomized into this arm. They may be provided with any combination of nutritional recommendations and supplements. Participants may need to use a mobile app in order to participate in the trial.
  Interventions: Dietary Supplement: VIOME-designed condition-based supplements

INTERVENTIONS:
Combination Product: VIOME Precision Nutrition Program — Precision supplement based on the participants microbiome sample results. Participants in this arm may have any combination of supplements, diet recommendations, and/or coaching.
  Other Names: VPNP
  Arms: Viome's Precision Nutrition Program
Dietary Supplement: VIOME-designed condition-based supplements — Pre-formulated supplements based on overall health conditions. Participants in this arm may have any combination of supplements, diet recommendations, and/or coaching.
  Other Names: VCS
  Arms: Viome's condition-based supplements

SUMMARY:
US residents who have gastrointestinal issues sign the informed consent form and are screened and enrolled for this study. Participants who are enrolled complete a survey upon enrollment and are randomized into one of three arms. This study is direct to participant and will NOT utilize clinical sites.

DETAILED DESCRIPTION:
Participants who meet the eligibility criteria are randomized into any of the three arms including: the control arm, VIOME's condition-based supplements (VCS) arm or the VIOME Precision Nutrition Program (VPNP) arm.

Placebo, Viome-designed condition-based supplements and Viome's Precision Nutrition Program include supplements, may include dietary recommendations towards improving the symptoms associated with gastrointestinal wellness. The trial will last approximately 4 months for each participant.

ELIGIBILITY:
Inclusion Criteria

* Resident of the United States
* Females and males ages 25-75 (inclusive)
* Able to speak and read English
* No unexplained weight loss, fevers, anemia, or blood in stool
* Willing and able to follow the trial instructions, as described in the recruitment letter
* Signed and dated informed consent prior to any trial-specific procedures.
* Diagnosis of IBS according to ROME IV criteria AND IBS-SSS score of 125-450 (inclusive)

Exclusion criteria

* Unwilling to change current diet
* Prior use of Viome products or services
* Antibiotic use in the previous 4 weeks
* Women who are pregnant (current or planned in the next 4 months), or breastfeeding
* < 90 days postpartum
* Active infection
* Unable or unwilling to use Viome's App on an iPhone or Android smartphone
* Significant diet or lifestyle changes in the previous 1 month
* IBD diagnosis
* Use of investigational drugs, products or devices within 1 month prior to and 4 months after the start of the trial
* Cancer therapy within the previous 1 year
* Major surgery in the last 6 months or planned in the next 4 months
* Prescribed any drug(s) that may interact with the supplement formulations
* Have any medical condition or allergy that may interact with, or prevents the healthy consumption of the supplements
* Allergies to any study-specific supplement ingredients
* Currently on a specific diet:

FODMAP KETO PALEO

- Gastrointestinal disease including: Esophagitis Celiac disease GI malignancy or obstruction Peptic ulcer Duodenal or gastric ulcer disease

* GI surgery except:

Appendectomy and benign polypectomy

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of VIOME's designed condition based supplements (VCS) | ~4 months
  Number of participants that show an improvement in GI health compared to baseline survey assessment.
Efficacy of VIOME Precision Nutrition Program (VPNP) | ~4months
  Number of participants that show an improvement in GI health compared to baseline survey assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, Principal Investigator — Viome
Locations (1):
- Viome Life Sciences, Bothell, Washington, United States